CLINICAL TRIAL: NCT01030484
Title: Nonalcoholic Fatty Liver Disease (NAFLD) Adult Database 2
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: NAFLD Adult Database 2 (IND); U01DK061730 (NIH)
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Liver Disease
Keywords: NAFLD; NASH; non-alcoholic steatohepatitis; fatty liver disease
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, liver tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NAFLD: adult patients with non-alcoholic fatty liver disease (NAFLD).

SUMMARY:
The NAFLD Database 2 will recruit at least 1,500 new adult participants suspected or known to have NAFLD or nonalcoholic steatohepatitis (NASH)-related cirrhosis and will also invite adult participants from the prior NAFLD Database and related studies (PIVENS trial and TONIC trial) to enroll in the NAFLD Database 2. To elucidate, through the cooperative effort of a multidisciplinary and multicenter group of collaborators, the etiology, natural history, diagnosis, treatment, and prevention of NAFLD, and in particular its more severe form of NASH and its complications.

DETAILED DESCRIPTION:
To add to the existing NAFLD Database an additional 1,500 adult participants with a diagnosis of NAFLD, supported by a recent liver biopsy, with a broad range of severity. Core data collection will include clinical, demographic, laboratory, imaging, and histological features

* To increase the population diversity of the NAFLD Database to provide greater representation of Hispanic, Native American, African American, and Asian patients among the new adult participants recruited into the NAFLD Database 2
* To expand the current specimen bank comprised of liver tissue, serum, plasma, and DNA obtained from new participants and continuing participants undergoing repeat liver biopsy with the specific goal of optimizing the collection of plasma or serum suitable for biomarker development studies by obtaining specimens in close temporal proximity to the performance of liver biopsy

ELIGIBILITY:
Inclusion Criteria:

Continuing participants:

* Previously enrolled in the NAFLD Database study, PIVENS or TONIC trials
* Age at least 18 years during the consent process
* Willingness to continue to be followed for up to 4 years
* Ability and willingness to give written, informed consent to be enrolled into Database 2

New participants:

* Age at least 18 years during the consent process
* Willingness to be followed for up to 4 years
* Ability and willingness to give written, informed consent to be screened for and, if eligible, to be enrolled into the Database 2 study
* Minimal or no alcohol use history consistent with NAFLD (see exclusion criteria)
* Collection of a standard of care liver biopsy that is obtained within 120 days of enrollment
* Collection of biosamples (serum, plasma, DNA, and, if available, liver tissue) within 90 days prior to enrollment and 0-90 days before or 4-90 days after the standard of care liver biopsy

Exclusion Criteria:

* Any condition or circumstances, which, in the opinion of the investigator, would interfere with completion of scheduled follow-up visits and procedures for the duration of the Database 2 study

  * Clinical or histological evidence of alcoholic liver disease: Regular and excessive use of alcohol within the 2 years prior to interview defined as alcohol intake greater than 14 drinks per week in a man or greater than 7 drinks per week in a woman. Approximately 10 g of alcohol equals one 'drink' unit. One unit equals 1 ounce of distilled spirits, one 12-oz beer, or one 4-oz glass of wine
  * Total parenteral nutrition for more than 1 month within a 6 month period before baseline liver biopsy
  * Short bowel syndrome
  * History of gastric or jejunoileal bypass preceding the diagnosis of NAFLD. Bariatric surgery performed following enrollment is not exclusionary. Liver biopsies obtained during bariatric surgery cannot be used for enrollment because of the associated surgical or anesthetic acute changes and the weight loss efforts that precede bariatric surgery
  * History of biliopancreatic diversion
  * Evidence of advanced liver disease defined as a Child-Pugh-Turcotte score equal to or greater than 10
  * Evidence of chronic hepatitis B as marked by the presence of HBsAg in serum (participants with isolated antibody to hepatitis B core antigen, anti-HBc total, are not excluded)
  * Evidence of chronic hepatitis C as marked by the presence of anti-HCV or HCV RNA in serum
  * Low alpha-1-antitrypsin level and ZZ phenotype (both determined at the discretion of the investigator)
  * Wilson's disease
  * Known glycogen storage disease
  * Known dysbetalipoproteinemia
  * Known phenotypic hemochromatosis (HII greater than 1.9 or removal of more than 4 g of iron by phlebotomy)
  * Prominent bile duct injury (florid duct lesions or periductal sclerosis) or bile duct paucity
  * Chronic cholestasis
  * Vascular lesions (vasculitis, cardiac sclerosis, acute or chronic Budd-Chiari, hepatoportal sclerosis, peliosis)
  * Iron overload greater than 3+
  * Zones of confluent necrosis, infarction, massive or sub-massive, pan-acinar necrosis
  * Multiple epithelioid granulomas
  * Congenital hepatic fibrosis
  * Polycystic liver disease
  * Other metabolic or congenital liver disease
  * Evidence of systemic infectious disease
  * Known HIV positive
  * Disseminated or advanced malignancy
  * Concomitant severe underlying systemic illness that in the opinion of the investigator would interfere with completion of follow-up
  * Active drug use or dependence that, in the opinion of the study investigator, would interfere with adherence to study requirements
  * Any other condition, which in the opinion of the investigator would impede compliance or hinder completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with suspected or known non-alcoholic fatty liver disease (NAFLD) or nonalcoholic steatohepatitis (NASH)-related cirrhosis of the liver
Sampling Method: Non-Probability Sample
Enrollment: 2501 (Actual)
Dates: Start 2009-12-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Liver histology scores | varies
  Liver histology scores (derived from central reading of liver biopsy at entry, standard of care biopsy done during screening or follow-up, or liver biopsy obtained for PIVENS or TONIC trials)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (8):
- United States (8):
  - University of California, San Diego, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Sanyal AJ, Van Natta ML, Clark J, Neuschwander-Tetri BA, Diehl A, Dasarathy S, Loomba R, Chalasani N, Kowdley K, Hameed B, Wilson LA, Yates KP, Belt P, Lazo M, Kleiner DE, Behling C, Tonascia J; NASH Clinical Research Network (CRN). Prospective Study of Outcomes in Adults with Nonalcoholic Fatty Liver Disease. N Engl J Med. 2021 Oct 21;385(17):1559-1569. doi: 10.1056/NEJMoa2029349. PMID 34670043
- [Derived] Vilar-Gomez E, Gawrieh S, Liang T, McIntyre AD, Hegele RA, Chalasani N. Interrogation of selected genes influencing serum LDL-Cholesterol levels in patients with well characterized NAFLD. J Clin Lipidol. 2021 Mar-Apr;15(2):275-291. doi: 10.1016/j.jacl.2020.12.010. Epub 2020 Dec 27. PMID 33454241
- See also: Nonalcoholic Steatohepatitis Clinical Research Consortium — http://jhuccs1.us/nash/
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/